CLINICAL TRIAL: NCT01989403
Title: The Long-term Course of Patients Undergoing Alternative and Integrative Therapy for Lumbar Disk Herniation: A Prospective Observational Study
Brief Title: Alternative and Integrative Therapy for Lumbar Disk Herniation
Status: Completed | Type: Observational
Sponsor: Jaseng Hospital of Korean Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: JS-CT-2011-03
Record Dates: First submitted 2013-11-04; First posted 2013-11-21 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Sciatica; Intervertebral Disc Disorder
MeSH Terms: conditions — Sciatica; Intervertebral disc disease | interventions — Phytotherapy; Acupuncture Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lumbar disc herniation patients: LBP with sciatica, with a numeral rating scale (NRS) leg pain intensity of 5 or higher and onset within 1 year; (2) LDH confirmed by MRI
  Interventions: Other: herbal medicine, acupuncture, bee-venom acupuncture, and Chuna manipulation

INTERVENTIONS:
Other: herbal medicine, acupuncture, bee-venom acupuncture, and Chuna manipulation

SUMMARY:
The investigators report management of lumbar disc herniation with severe sciatic pain using an integrative complementary and alternative medicine approach with a 5 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* LBP with sciatica,
* A numeral rating scale (NRS) leg pain intensity of 5 or higher
* Onset within 1 year;
* Lumbar Disk Heriation confirmed by MRI;
* Written consent to attend 6 months of integrative CAM treatment and following assessment visits.

Exclusion Criteria:

* Treatment regarding the current LBP and/or sciatica (e.g. surgery, nerve block, or analgesic medication) other than the CAM treatment specified in the protocol
* Non-spinal or soft tissue problem related to back pain or sciatica (e.g. pregnancy, spinal tumor, or rheumatoid arthritis)
* History of spinal surgery, vertebral dislocation, fracture, or cancer;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: integrative hospital that offers both Western and traditional Korean medical services
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale for low back and leg pain | Changes from Baseline in Visual analogue scale at 2 weeks, 4 weeks, 8weeks, 12weeks, 20weeks, 24weeks, 1 years, 2years,3years,4years and 5years.
the Oswestry Disability Index | Changes from Baseline in the Oswestry Disability Index at 2 weeks, 4 weeks, 8weeks, 12weeks, 20weeks, 24weeks, 1 years, 2years,3years,4years and 5years.
the SF-36 Health Survey | Changes from Baseline in the SF-36 Health Survey at 2 weeks, 4 weeks, 8weeks, 12weeks, 20weeks, 24weeks, 1 years, 2years,3years,4years and 5years.

SECONDARY OUTCOMES:
Straight Leg Raise test | Changes from Baseline in the Straight Leg Raise test at 2 weeks, 4 weeks, 8weeks, 12weeks, 20weeks, 24weeks, 1 years, 2years,3years,4years and 5years.
Adverse events | at 2 weeks, 4 weeks, 8weeks, 12weeks, 20weeks, 24weeks, 1 years, 2years,3years,4years and 5years.
  Skin and general reactions, aggravation or change in pain before and after acupuncture, pharmacoacupuncture, and Chuna manipulation treatment were observed.
  Regular blood tests (blood cell count, liver, renal function tests, inflammatory activity indexes) were administered.

CONTACTS AND LOCATIONS:
Locations (1):
- Jaseng Spine and joint Research Institute, Seoul, South Korea